CLINICAL TRIAL: NCT02042014
Title: An Open-label, Multi-center Protocol to Provide QTI571 to PAH Patients Who Participated in the Extension Study (A2301E1) in Japan and Are Judged by the Investigator to Benefit From Continued QTI571 Treatment
Brief Title: Open-label, Multi-center Protocol to Provide QTI571 to PAH Patients Who Participated in the Extension Study (A2301E1) in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQTI571AJP01
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Severe Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension, QTI571, open label study
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: This was a multi-center open label study to provide continued supply of QTI571 to patients in Japan who were treated in the extension study (A2301E1) and were judged by the investigator to benefit from continued QTI571 treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QTI571 (Experimental): Participants will receive QTI571 during 3 years.
  Interventions: Drug: QTI571

INTERVENTIONS:
Drug: QTI571 — QTI571 200mg up to 400mg (depending on tolerability) taken orally, once a day.

SUMMARY:
To provide continued treatment to Pulmonary Arterial Hypertension (PAH) patients who are benefitting from treatment with QTI571.

DETAILED DESCRIPTION:
This was a multi-center open label study to provide continued supply of QTI571 to patients in Japan who were treated in the extension study (A2301E1) and were judged by the investigator to benefit from continued QTI571 treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient is receiving QTI571 for the treatment of Pulmonary Arterial Hypertension (PAH) and is currectly enrolled in a long-term extension study (CQTI571A2301E1) in Japan.
* Patient is currently benifitting form the treatment with QTI571 in the opinion of the investigator.

Exclusion Criteria:

* Patient has been permanently discontinued from QTI571 study treatment in the parent study.
* Concomitant use of oral vitamin K antagonist medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 participants entered this study after completing the CQTI571A2301E1 study. All 8 participants discontinued study prematurely.
Groups:
- QTI571: Participants received QTI571 during 3 years
Period: Overall Study
Arm/Group | QTI571
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Physician Decision | 7

BASELINE CHARACTERISTICS:
Arm/Group | QTI571
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: All Serious Adverse Events were evaluated and reported for all participants receiving QTI571. 16 individual SAEs were observed in 5 subjects.
Time Frame: Approximately 2.9 years
Measure: Number; unit: participants
Arm/Group | QTI571
Number analyzed (Participants) | 8
participants
  Cardiac disorders (5 events) | 5
  Infections and infestations (5 events) | 3
  Resp, thoracic,mediastinal & disorder (2 events) | 1
  Product issues (3 events) | 1
  Death (none) | 0
  Skin & subcutaneous tissue disorder(1 event) | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to approximately 2.9 years
Description: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 2.9 years. All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 2.9 years
Groups:
- QTI571: QTI571
Arm/Group | QTI571
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QTI571 (N=8)
Acute myocardial infarction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 3
Supraventricular tachycardia (Cardiac disorders) | 1
Cellulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Device connection issue (Product Issues) | 1
Device occlusion (Product Issues) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
No efficacy data was captured in this study, and no analysis of efficacy was planned. No formal analyses of Adverse Events were undertaken.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.